CLINICAL TRIAL: NCT01205802
Title: Prospective Study on Usability of Ringed Polytetrafluoroethylene Graft for Venous Vascular Reconstruction of Living Donor Liver Transplantation
Brief Title: Usability of Ringed Polytetrafluoroethylene Graft for Venous Vascular Reconstruction of Living Donor Liver Transplantation
Acronym: MHVLDLT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Asan Medical Center (Other)
Responsible Party: Shin Hwang / Professor, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHV_Goretex_LDLT
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Patency, Hepatic Venous Congestion
Keywords: patency, hepatic venous congestion, liver transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTFE group (Active Comparator): MHV reconstruction with ringed Goretex
  Interventions: Procedure: MHV reconstruction
- Homograft group (Placebo Comparator): MHV reconstruction with homograft
  Interventions: Procedure: MHV reconstruction

INTERVENTIONS:
Procedure: MHV reconstruction — MHV reconstruction with PTFE or homograft

SUMMARY:
Middle hepatic vein (MHV) reconstruction with an interposition vessel graft has been settled as a standard procedure for living donor liver transplantation (LDLT) using a right lobe graft. Increasing demand of vessel graft in the situation of limited resources of allograft led the investigators to search for new vessel substitutes. Since the use of thin-walled expanded polytetrafluoroethylene (PTFE) graft showed poor long-term patency, a prospective study is going to be performed to enhance the clinical usability of expanded PTFE graft. A clinical study intends to know how to maintain its luminal flow effectively by using ringed PTFE graft. During 12 months of study period, ringed PTFE graft will be used for reconstruction of MHV reconstruction. The investigators expect that ringed PTFE graft seems to be a more useful alternative than usual PTFE graft when adequate autologous or allogenic vessel graft is not available.

DETAILED DESCRIPTION:
Since late 2009, the relative supply of vessel allograft over the increasing demand on LDLT became seriously shortened in the investigators' institution. Thus the investigators decide to use prosthetic vascular grafts more frequently than before. After a preliminary study from January 2010 to July 2010, a prospective case-controlled study will be performed for 12 months from August 2010 to July 2011.

The case number of patients requiring MHV reconstruction is expected as being 200 during the study period. Of them, currently using homologous or autologous vessel grafts will be used for 150. Due to expected shortage of such human vessels, other 50 will undergo MHV reconstruction using ringed PTFE graft in addition to available autologous or homologous vessel segments.

According to the implications from precedent animal and preliminary studies, the investigators set up the institutional guidelines for use of prosthetic vascular graft during MHV reconstruction of LDLT as follows: use only ringed PTFE graft; choose graft of a larger-caliber (≥1 cm); apply an intervening patch when making an end-to-side anastomosis for MHV branch of the segment 8 (V8); provide a slight redundancy in length; make the IVC-side orifice much larger than the usual; perform flow surveillance more frequently with dynamic CT scan and Doppler ultrasonography; place a stent as soon as any significant luminal narrowing is detected; and keep hypocoagulable state for at least 2 weeks and anti-platelet therapy for 6 months.

Technical knacks for secure suture include minimal removal of the rings attached at the surface of the ringed PTFE, use of PTFE suture material (GORE-TEX SUTURE; GORE-TEX, W.L. Gore & Associated, Inc., USA) - a non-absorbable monofilament made of expanded PTFE enabling 1:1 needle to thread ratio to minimize needle hole bleeding at anastomoses, making a redundant patch plasty for end-to-side branch anastomosis especially for V8, and spray application of fibrin glues for suture-point minute bleedings and for stable fixation of PTFE graft at the liver cut surface.

The primary goal for this clinical study is set to keep up the rate of luminal patency as 100% for at least 1 month after MHV reconstruction for LDLT. Any occurrence of flow disturbance at luminal narrowing greater than 50% of the original cross-sectional area at 1 month should make the guidelines revise extensively. This protocol is designed as being a prospective case-controlled study for 1 year.

The use of PTFE graft for various hepatobiliary surgical procedures including LDLT has been permissible in the investigators' institution. Only after parenchymal transection of the donor liver, the size and shape of suitable vessel allograft for MHV reconstruction is determined. Thus the use of PTFE graft will be decided at this time after checking the list of all available allograft stored at the institutional tissue bank. The indication of PTFE use will be confined to the occasions that adequate allograft was not available. Permission for potential use of PTFE graft will be obtained from all cases of LDLT using a right lobe graft. This study protocol is approved by the institutional review board for clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Living donor liver transplantation requiring MHV reconstruction

Exclusion Criteria:

* Living donor liver transplantation not requiring MHV reconstruction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Patency of the reconstructed MHV | Follow-up for 1 year
  Patency rate up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Hwang S, Jung DH, Ha TY, Ahn CS, Moon DB, Kim KH, Song GW, Park GC, Jung SW, Yoon SY, Namgoong JM, Park CS, Park YH, Park HW, Lee HJ, Lee SG. Usability of ringed polytetrafluoroethylene grafts for middle hepatic vein reconstruction during living donor liver transplantation. Liver Transpl. 2012 Aug;18(8):955-65. doi: 10.1002/lt.23456. PMID 22511404